CLINICAL TRIAL: NCT01008241
Title: Project Hope: Survey of South Florida Residents Knowledge and Opinions on End-of-Life Issues
Brief Title: South Florida Residents Knowledge and Opinions on End-of-Life Issues
Status: Completed | Type: Observational
Sponsor: Maria Isabel Fernandez (Other)
Responsible Party: Sponsor-Investigator, Maria Isabel Fernandez, Pre-Doctoral Behavioral Research Fellow College of Osteopathic Medicine, Nova Southeastern University
Organization: Nova Southeastern University (Other)
Other Study IDs: Project Hope
Record Dates: First submitted 2009-11-03; First posted 2009-11-05 (Estimated); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Death
Keywords: Hospice; End of Life; Knowledge; Attitudes; Opinions; Advanced Care Planning; Death and Dying; Communication
MeSH Terms: conditions — Death; Behavior; Communication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Group: Convenience sample of adult residents of South Florida
  Interventions: Behavioral: Paper questionnaire

INTERVENTIONS:
Behavioral: Paper questionnaire — Participants will complete a paper and pencil questionnaire that measures 4 domains of interest (advanced care planning; end of life care; hospice care and death and dying) as well as demographic factors (age, marital status, education etc.)

SUMMARY:
The goal of this cross-sectional study is to gain an understanding of the knowledge and attitudes regarding end of life issues and hospice care among a sample of residents of South Florida. This study is being conducted by 3rd year Osteopathic Medical Student (OMS-III)Nova Southeastern University College of Osteopathic Medicine (NSU COM) research fellow Heather Ruff as part of the research fellowship requirements.

Participants will complete a paper and pencil questionnaire that measures 4 domains of interest (advanced care planning; end of life care; hospice care and death and dying) as well as demographic factors (age, marital status, education etc.). It is estimated that the survey will take 15 minutes to complete. Data will be collected anonymously, with no personal identifying information. The instructions on the questionnaire state that by completing the questionnaire, the participant is providing consent to participate in the study. We will use time and space sampling methods to recruit up to 250 participants at community venues (i.e., beaches, street corners, parks, pedestrian malls, and other public venues were people congregate) in South Florida. At each venue, we will define a specific area; persons who enter the defined area will be approached, screened for eligibility (18 years of age or older and a resident of South Florida), and if eligible, invited to participate by trained research staff. Sampling intervals will be determined by traffic flow at each venue. If a person agrees to participate they will be given a paper and pencil copy of the survey to complete on the spot. Participants will be given a token of appreciation. Data entry and data analyses will be done using Statistical Package for the Social Sciences (SPSS).

DETAILED DESCRIPTION:
The survey instrument included questions about demographics (constructed by the researchers), including the participants' age, gender, ethnicity, relationship status, education level, income, and whether they had a religious affiliation. Also included were items about steps participants may have taken to plan for their health care in the event they were unable to make personal health care decisions, such as whether they had a living well or durable power of attorney for health care, and whether they had knowledge of the existence of these documents prior to taking the survey. Participants were also asked where/from whom they first learned about hospice and where they got most of their knowledge about hospice. Hospice. This scale contained 24 statements about knowledge and opinions on hospice care. Hospice was defined as a program that provides care to people with illnesses that cannot be cured when they are at the end of their lives. Participants were asked to report their feelings from 1 (strongly disagree) to 5 (strongly agree) about each statement. Items included (a) ''Hospice care means giving up,'' (b) ''Hospice care means you get no treatment,'' (c) ''Hospice care can be provided in a patient's home if the patient or family wishes it,'' and (d) ''Those who believe in God do not need hospice.'' More favorable attitudes toward hospice are evidenced in higher scores. End of life care. Seven Likert-type items were used to ask participants about their thoughts and feelings related to the kind of medical care they would want if they had a disease, like cancer, that could not be cured. When answering these questions, participants were asked to consider a hypothetical situation in which they had a terminal disease and not consider their current state of health. This scale is composed of 7 items and uses a 5-point Likert-type response ranging from 1 (strongly disagree) to 5 (strongly agree). Participants were asked items such as

(a) ''If I had a disease (like cancer) that the doctors could not cure, I would want to live as long as possible even if I had to be on life support or a breathingmachine,'' and (b) ''If I had a disease (like cancer) that could not be cured, decreasing pain would be more important to me than living as long as possible.'' Higher scores indicate higher levels of advanced planning for EOL care. Communication about death and dying. Death and dying communication was measured using 9 items rated on a 5-point Likert format, with responses ranging from 1 (strongly disagree) to 5 (strongly agree). Examples of items include

1. ''I feel comfortable talking about death in general,''
2. ''Dying is a normal part of life,'' and (c) ''Death should be avoided at all costs.'' Higher scores indicate greater comfort with communicating about death and dying. Through convenience sampling strategies, a total of 625 individuals were approached; 610 were eligible, and 361 participants returned the survey. Thirty questionnaires were dropped because less than two thirds of the scale items were completed), resulting in a sample size of 331. Due to low numbers in some demographic categories, educational level was collapsed into 3 categories (ie, high school/some college, associate/ bachelors degree, and graduate degree) and annual income was collapsed into ''less than US$25 000, $25 000 to US$49 999, and US$50 000 or more. Ethnicity was categorized as non-Hispanic white, black, Hispanic, and other/mixed race. Relationship status was dichotomized into ''have a partner'' and ''do not have a partner.''

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* Resident of Broward or Miami-Dade counties

Exclusion Criteria:

* Less than 18 years of age
* Not currently residing in Broward or Miami-Dade counties

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult residents of South Florida
Sampling Method: Non-Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
attitudes towards end of life issues | one time point
  brief attitude scale to document perceptions of end of life issues

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Ruff, B.S., Principal Investigator — Nova Southeastern University College of Osteopathic Medicine; Maria I Fernandez, Ph.D., Study Chair — Nova Southeastern University College of Osteopathic Medicine; Stephen Bowen, M.D., M.P.H., Study Chair — Nova Southeastern University College of Osteopathic Medicine; Robin J Jacobs, Ph.D., Study Chair — Nova Southeastern University College of Osteopathic Medicine; Hilary Gerber, B.S., Study Chair — Nova Southeastern University College of Osteopathic Medicine
Locations (2):
- United States (2):
  - A variety of public venues in Broward County, Fort Lauderdale, Florida
  - A variety of public venues in Miami-Dade County, Miami, Florida